CLINICAL TRIAL: NCT05782829
Title: Perioperative Stress Management in Outpatient Surgery With L-tyrosine Supplementation
Brief Title: Perioperative Stress Management in Outpatient Surgery With L-tyrosine Supplementation (SPOT)
Acronym: SPOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-16
Record Dates: First submitted 2023-02-13; First posted 2023-03-24 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Stress
Keywords: L-Tyrosine supplementation; Perioperative stress

STUDY DESIGN:
Intervention Model Description: prospective, monocentric, double-blind randomized study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-Tyrosine (Experimental)
  Interventions: Dietary Supplement: L-tyrosine supplementation
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo supplementation

INTERVENTIONS:
Dietary Supplement: L-tyrosine supplementation — L-Tyrosine supplementation before surgery for inguinal hernia under general anaesthesia
  Arms: L-Tyrosine
Dietary Supplement: Placebo supplementation — Placebo supplementation before surgery for inguinal hernia under general anaesthesia
  Arms: Placebo

SUMMARY:
Patient undergoing surgery is exposed to many stressors: diachronic (gesture anticipation), synchronic (intraoperative aggression) and historical (subject's personality). Reducing the level of stress experienced is a factor for improving the quality of the surgical gesture and the simplicity of the follow-up. The previous methods used were intended to reduce the body's reactivity to aggressions through anaesthesia consultation and L-Tyrosine supplementation. Currently with the progression of outpatient surgery and the need for early rehabilitation, L-Tyrosine supplementation is suppressed to improve recovery. Some patients, however, have a high level of stress that may require anxiolysis when the ideal treatment does not exist (ineffective hydroxyzine, benzodiazepines having many side effects). The strategy of this work is to improve the body's ability to respond to stressors, by administering l-tyrosine with no impact on waking or returning home.

ELIGIBILITY:
Inclusion Criteria:

* Membership of a social security scheme or equivalent
* At least 18 years of age
* Able to express consent
* Indication of unilateral or bilateral inguinal hernia cure
* General anaesthesia proposed and retained for inguinal hernia treatment regardless of surgical technique

Exclusion Criteria:

* Surgical indication for another reason or hernial cure associated with another procedure
* Smoking estimated at more than 35 pack-years
* History of psychiatric pathology
* ASA 3 or 4 according to the American Society of Anesthesiologists classification. As a reminder, an ASA 3 class concerns a patient with a severe but not disabling general disease, and an ASA 4 class concerns a patient with a disabling general disease involving the vital prognosis.
* ASA 2 and having at least one of the following pathologies or patients treated with -blockers: insulin-dependent diabetes, high blood pressure, heart rhythm disorder, dysthyroidism, progressive neurological disease, long-term benzodiazepines.
* Starch allergy or intolerance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Variation of anxiety status | between the day before surgery and thes day after surgery
  Anxiety score measured using Y-A STAI

SECONDARY OUTCOMES:
Other stress markers variation | the day before surgery
  anxiety visual analogue scale (from 0 to 10, 10 is worst)
Other stress markers variation | the day after surgery
  anxiety visual analogue scale (from 0 to 10, 10 is worst)
Other stress markers variation | the day before surgery
  heart blood pressure (Systolic and diastolic)
Other stress markers variation | the day after surgery
  heart blood pressure (Systolic and diastolic)
Other stress markers variation | the day before surgery
  cortisol dosage
Other stress markers variation | the day after surgery
  cortisol dosage

CONTACTS AND LOCATIONS:
Locations (1):
- CHPG, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No
Not scheduled